CLINICAL TRIAL: NCT01889836
Title: Brazil's Conjugated Vaccine Project Against Meningococcal C. Safety and Immunogenicity Study in Young Adults the Meningococcal Serogroup C Vaccine Produced by Bio-Manguinhos
Brief Title: Safety and Immunogenicity Study in Young Adults the Meningococcal Serogroup C Vaccine Produced by Bio-Manguinhos
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASCLIN / 001 / 2013
Record Dates: First submitted 2013-06-10; First posted 2013-07-01 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Meningitis, Meningococcal, Serogroup C
Keywords: meningococcal conjugate vaccine serogroup C; Prevention
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MenCC-Bio (Experimental): The experimental group will receive one dose of meningococcal C vaccine adsorbed produced by Bio-Manguinhos.
  Interventions: Biological: 'MenCC-Bio'
- MENJUGATE® (Active Comparator): The control group will receive one dose of meningococcal C vaccine adsorbed - MENJUGATE®.
  Interventions: Biological: MENJUGATE

INTERVENTIONS:
Biological: 'MenCC-Bio' — The experimental group will receive one dose of meningococcal C vaccine adsorbed produced by Bio-Manguinhos.
  Arms: MenCC-Bio
Biological: MENJUGATE — The control group will receive one dose of meningococcal C vaccine adsorbed - MENJUGATE.
  Arms: MENJUGATE®

SUMMARY:
Clinical trial phase I, randomized, double blind, where 30 individuals will receive the experimental vaccine while 30 other volunteers will receive a meningococcal C conjugate vaccine already licensed in Brazil and available in the National Immunization Program for children less than 12 months of age. The primary outcome of the study is to evaluate the safety profile of the vaccine under test, which should allow its application in humans. Secondly, the investigators will study its immunogenicity from the evaluation of the correlates of seroprotection for meningococcal, defined by the World Health Organization (WHO).

DETAILED DESCRIPTION:
Study design - This is a clinical study Phase I, randomized, double blind with 60 individuals. 30 individuals will receive the experimental vaccine by Bio-Manguinhos/Fiocruz and 30 individuals will receive a meningococcal C conjugated vaccine used in the National Immunization Program.

Location of Study - Clinical Trials Unit for Immunobiology by Bio-Manguinhos/Fiocruz.

Primary objective - Evaluate the safety of the meningococcal C vaccine by Bio-Manguinhos/Fiocruz for use in humans.

Secondary objective - To evaluate the immunogenicity of the meningococcal C vaccine by Bio-Manguinhos in young adults.

specific objectives

1. To evaluate the frequency / intensity of adverse events occurring up to 30 days after vaccination.
2. To evaluate the seroconversion defined as pre-immunization serum nonreactive (negative) and post-immunization reactor (positive) antigens, with getting titles 8 (rabbit complement) to the target strain used in the test of bactericidal power of the sera from immunized volunteers, a 4-fold increase in titers following vaccination compared to pre-vaccination and antibody titers after immunization.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Age between 18 and 50.
* Available for follow-up during the period of the study
* Willing to provide their name, address, telephone number and other information by each they can be contact for the study learn if necessary (eg in case of lack the scheduled visit).
* Willing to strictly follow the study protocol.
* Ability to understand and signing the consent form.
* Understanding the impossibility to participate in another clinical trial during the time which is participating in the study.
* Intellectual level that allows filling in the forms for registration of symptoms at home.
* Acceptance for serological testing for human immunodeficiency virus (HIV), Hepatitis B virus (HBV) and Hepatitis C virus (HCV).
* Be in good health, with no significant medical history.
* Physical examination screening without significant clinical changes.
* Screening laboratory tests within normal limits established the laboratory or abnormal values smaller than 1 degree.
* Additional criterion for females: Negative pregnancy test before application of the vaccine dose, for women of childbearing age.

Exclusion Criteria:

- Pregnant or breast-feeding.

Personal history of:

* Meningitis of any kind.
* Serious adverse reaction to any vaccination, such as difficulty breathing, angioedema and anaphylaxis.
* Severe adverse reaction related to prior immunization with tetanus and / or diphtheria vaccines alone or in combination vaccines.
* Vaccination with tetanus and diphtheria vaccines alone or in combinations vaccine in the last two years.
* Use of allergy shots antigens within 14 days or less prior to vaccination.
* Immunoglobulin in the last 12 months before vaccination.
* Use of blood products in the last 12 months before vaccination.
* Use of any vaccine 30 days before vaccination.
* Chronic use of any medication except homeopathic and trivial as Nasal saline and vitamins.
* Previous use of cytotoxic or immunosuppressive medication. Are acceptable individuals who have made use of this type of immunosuppressive medication in doses not more than six months, such as nasal steroids for allergic rhinitis or dermatitis to topical corticosteroid uncomplicated.
* Use of any investigational medication over a period of 1 year prior to vaccination.
* Unstable asthma or has required urgent care, hospitalization or intubation in the last two years, or requiring use of oral or intravenous corticosteroids.
* Severe anaphylaxis or angioedema.
* Neurological, cardiovascular, respiratory, hepatic, renal, hematologic, rheumatologic or autoimmune clinically significant (diseases that have led to hospitalization or prolonged treatment).
* Coagulopathy diagnosed by a medical report or capillary fragility (eg bruising or bleeding without justifiable cause).
* Seizures, except that they have been fever, before 2 years of age.
* Psychiatric illness that impairs adherence to protocol, such as psychoses, neuroses obsessive-compulsive disorder, bipolar disorder being treated, diseases requiring lithium treatment and suicidal ideation in the last five years prior to enrollment.
* Active malignancy (eg any type of cancer) or treated to recourse during the study.
* Sickle cell anemia.
* Asplenia (or absence of spleen removal of same).
* HIV positive in the screening test or history of any immunosuppressive disease.
* Positive serology for hepatitis C screening test.
* HBsAg positive in the screening test.
* Alcoholism (CAGE criterion), used for detection of abusive drinkers and alcoholics, validated in our population with a sensitivity of 88% and specificity of 83% if two or more responses among four possible, are affirmative.
* Use / abuse of drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the meningococcal C vaccine by Bio-Manguinhos/Fiocruz for use in humans. | Adverse events post vaccination will be evaluated on days 1,3, 10 and 15 by phone call and on days 2, 7 and 30 at the research center
  To evaluate the frequency / intensity of adverse events occurring up to 30 days after vaccination.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the meningococcal C vaccine by Bio-Manguinhos in young adults. | Blood collection 30 days after vaccination
  30 days after vaccination, blood sampling will be conducted which composes for serological analysis of immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Guimarães de Noronha, MsD, Principal Investigator — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz)
Locations (1):
- Unidade de Ensaios Clínicos para Imunobiológicos, Rio de Janeiro, Rio de janeiro/RJ, Brazil